CLINICAL TRIAL: NCT02518984
Title: Atrial Fibrillation General Long Term Registry
Brief Title: Atrial Fibrillation General Registry
Acronym: AFGenLT
Status: Completed | Type: Observational
Sponsor: European Society of Cardiology (Network)
Responsible Party: Sponsor
Other Study IDs: AFGen Long Term
Record Dates: First submitted 2015-04-16; First posted 2015-08-10 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Given the advances in Atrial Fibrillation (AF) management and the availability of new European Society of Cardiology (ESC) guidelines, there is a need for the systematic collection of contemporary data regarding the management and treatment of AF in the member ESC countries. It is now nearly 10 years since the last European registry of AF management was undertaken (as part of the ESC Euro Heart Survey programme), and a new registry was needed.

DETAILED DESCRIPTION:
Given the advances in Atrial Fibrillation (AF) management and the availability of new European Society of Cardiology (ESC) guidelines, there is a need for the systematic collection of contemporary data regarding the management and treatment of AF in the member ESC countries. It is now nearly 10 years since the last European registry of AF management was undertaken (as part of the ESC Euro Heart Survey programme), and a new registry was needed.

New guidelines on the management of AF have recently been published by the ESC, but it remains unclear how often clinicians adhere to them. Since the last Euro Heart survey, a change in management strategy has necessitated an update on prevalent management practices in AF. This is influenced by clinical availability of catheter ablation as a routine procedure and new antiarrhythmic drugs, and also by developments in stroke thromboprophylaxis and medical therapy options. Under the EURObservational Research Programme (EORP), an AF ablation sentinel pilot registry was launched in 2010.

A survey of AF management under the EORP programme will enable a timely assessment of the uptake of the new ESC guidelines, allow monitoring of implementation and uptake of catheter ablation, new antithrombotic drugs and new antiarrhythmic agents, and will inform about outcomes related to guideline-adherent management of AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be officially enrolled in the study only if ECG diagnosis of AF has been made.
* The qualifying episode of AF should have occurred within one year before the date of baseline.
* AF is the primary or secondary diagnosis, i.e. the current admission / visit may be due to other reasons.
* Patients need not be in AF at the time of enrolment.
* Signed Patient Inform Consent if applicable.

Exclusion Criteria:

* No ECG/Holter with AF recorded.
* Only atrial flutter recorded.
* The qualifying episode of AF occurred more than one year before the date of baseline.
* Age <18 years.
* Patients are already included in the ESC Atrial Fibrillation Long-Term registry if your centre was enrolled in the Pilot phase.
* Patients who are currently or are planned to be taking part in a cardiac clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out patients with AF and patients with acute pre-existing or new onset AF
Sampling Method: Non-Probability Sample
Enrollment: 19754 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
vital status | Baseline

OTHER OUTCOMES:
vital status | one year follow-up
vital status | two year follow-up
vital status | three year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Lip, MD, Study Chair — European Society of Cardiology
Locations (1):
- European Society of Cardiology, Biot, France

IPD SHARING:
Plan to Share IPD: No